CLINICAL TRIAL: NCT02951039
Title: Non-Interventional Study on Edoxaban Treatment in Routine Clinical Practice for Patients With Non Valvular Atrial Fibrillation (NVAF)
Brief Title: Edoxaban Treatment in Routine Clinical Practice for Patients With Atrial Fibrillation in Korea and Taiwan (ETNA-AF-KOR-TWN)
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DU176b-C-A4008
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation
Keywords: Non valvular Atrial Fibrillation; Non-interventional Study; Efficacy/Safety; Real World Evidence
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Edoxaban: Patients with established NVAF treated with edoxaban according to package information. Physician's prescribing behaviour will not be influenced; patients may only be included after the treating physician has made the clinical decision to prescribe edoxaban.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Prescribed according to approved label
  Other Names: Lixiana

SUMMARY:
In order to understand the risks and benefits of edoxaban use in a real-world clinical setting in the Non valvular Atrial Fibrillation (NVAF) indication, Daiichi-Sankyo proposed this non-interventional study to gain insight into the safety (bleeding, liver adverse events, all-cause mortality and other drug related adverse events) and efficacy of edoxaban use in non-preselected patients with NVAF.

DETAILED DESCRIPTION:
Edoxaban was approved by the Ministry of Food and Drug Safety (MFDS) in Korea (date: 25th, August 2015) for the reduction in the risk of stroke and systemic embolism in patients with NVAF, treatment of deep vein thrombosis (DVT) and pulmonary embolism. Edoxaban was approved by the Taiwan Food and Drug Administration (TFDA) in Taiwan (date: 24th, February, 2016) for the prevention of stroke and systemic embolism in adult patients with NVAF with one or more risk factors, such as congestive heart failure, hypertension, age at least 75 years, diabetes mellitus, prior stroke or transient ischemic attack (TIA), or treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE), following 5 to 10 days of initial therapy with a parenteral anticoagulant.

Real world evidence data of routine clinical practice use of edoxaban up to two years will be collected and evaluated in approximately 2,500 patients, treated by specialized as well as non-specialized physicians in hospital centers.

ELIGIBILITY:
Inclusion Criteria:

* NVAF-patients treated with edoxaban according to Summary of Product Characteristics (SmPC).
* Written informed consent for participation in the study (ICF).
* Not simultaneously participating in any interventional study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with NVAF and treated with edoxaban according to the package information.
Sampling Method: Non-Probability Sample
Enrollment: 3008 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Rate of Participants Experiencing Real-World Safety Data Events within 2 Years | within 2 years
  Real-world safety data events include bleeding events (including intracranial haemorrhage), adverse events and mortality

SECONDARY OUTCOMES:
Rate of Participants with Patient Relevant Outcomes | within 2 years
  Patient relevant outcomes include Strokes (ischaemic and haemorrhagic) , Systemic Embolic Events (SEE), Transient Ischemic Attack (TIA), Major Adverse Cardiovascular Events (MACE), Venous Thromboembolism (VTE), Acute Coronary Syndrome (ACS), and Hospitalisations related to a cardiovascular (CV) condition.
Rate of Participants Compliant with Edoxaban Therapy | 2 years
  Categories: Always, Almost Always, Most of the Time, Less than Half the Time, Unknown

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (47):
- South Korea (37):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - GangNeung Asan Hospital, Gangneung, Gangwon-do
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Samsung Changwon Hospital, Changwŏn, Gyeongsangnam-do
  - St. Carollo General Hospital, Suncheon, Jeollanam-do
  - Gyeongsang National University Hospital, Gyeongsang, Jinju-si
  - Inje Universitiy Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Dong A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeongnam University Medical Center (1526), Daegu
  - Yeongnam University Medical Center (1533), Daegu
  - Chungnam National University Hospital, Daejeon
  - Chosun University Hospital, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital (1512), Seoul
  - Seoul National University Hospital (1534), Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Veterans Health Service Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center (1519), Seoul
  - Samsung Medical Center (1520), Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Hallym University, Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Taiwan (10):
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - Chang Gung Memorial Hospital, Linko, Taoyuan District, Guishan District
  - Tri-Service General Hospital, Taipei, Neihu District
  - Chang Gung Memorial Hospital, KaoHsiung, Kaohsiung City, Niaosong District
  - Taichung Veterans General Hospitial, Kaohsiung City, Niaosong District
  - Cheng Hsin General Hospital, Taipei, Pai-Tou
  - National Taiwan University Hospital, Taipei, Zhongzheng District
  - KaoHsiung Veterans General Hospital, Kaohsiung City, Zuoying District
  - Chung Shan Medical University Hospitial, Taichung
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Derived] Morrone D, Dinshaw L, de Souza JAG, Chen C, Kirchhof P, Koretsune Y, Pecen L, Wang CC, Yamashita T, Unverdorben M, De Caterina R. Edoxaban treatment in routine clinical practice is highly concordant with the 2020 European Society of Cardiology atrial fibrillation guidelines: results from the noninterventional Global ETNA-AF programme. Eur Heart J Open. 2025 Mar 28;5(2):oeaf004. doi: 10.1093/ehjopen/oeaf004. eCollection 2025 Mar. PMID 40161305
- [Derived] De Caterina R, Unverdorben M, Chen C, Choi EK, Koretsune Y, Morrone D, Pecen L, Bramlage P, Wang CC, Yamashita T, Kirchhof P. Two-Year Follow-Up of Patients With Atrial Fibrillation Receiving Edoxaban in Routine Clinical Practice: Results From the Global ETNA-AF Program. Clin Cardiol. 2025 Feb;48(3):e70091. doi: 10.1002/clc.70091. PMID 40014354
- [Derived] Unverdorben M, Colonna P, Jin J, Kohler S, Santamaria A, Saxena M, Borrow A, Chen C, von Heymann C, Vanassche T. Periprocedural Edoxaban Management and Clinical Outcomes in Patients Undergoing Transcatheter Cardiovascular Procedures in the EMIT-AF/VTE Program. Clin Appl Thromb Hemost. 2024 Jan-Dec;30:10760296241260728. doi: 10.1177/10760296241260728. PMID 38881370
- [Derived] von Heymann C, Unverdorben M, Colonna P, Santamaria A, Saxena M, Vanassche T, Kohler S, Borrow AP, Jin J, Chen C. Management of edoxaban therapy and clinical outcomes in patients undergoing major or nonmajor surgery: a subanalysis of the EMIT-AF/VTE study. Thromb J. 2023 Dec 14;21(1):124. doi: 10.1186/s12959-023-00568-2. PMID 38098072